CLINICAL TRIAL: NCT02326558
Title: Comparison of Zero Ischemia Laparoscopic Microwave Ablation-Assisted Enucleation and Conventional Laparoscopic Partial Nephrectomy in the Treatment of T1a Renal Cell Carcinoma
Brief Title: Comparison of Microwave Ablation-Assisted Enucleation and Conventional Laparoscopic Partial Nephrectomy in the Treatment of T1a Renal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Huang Yi-Ran, Chef of Urology, RenJi Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-URO-001
Record Dates: First submitted 2014-12-17; First posted 2014-12-29 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Renal Cell Carcinoma
Keywords: zero ischemia; microwave; ablation; enucleation; renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- microwave enucleation (Experimental): zero ischemia laparoscopic microwave ablation-assisted enucleation of the tumor
  Interventions: Procedure: laparoscopic microwave ablation-assisted enucleation
- laparoscopic partial nephrectomy (Active Comparator): conventional laparoscopic partial nephrectomy with clamping of the renal artery
  Interventions: Procedure: conventional laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: laparoscopic microwave ablation-assisted enucleation
  Arms: microwave enucleation
Procedure: conventional laparoscopic partial nephrectomy
  Arms: laparoscopic partial nephrectomy

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety and efficiency of zero ischemia laparoscopic microwave ablation-assisted enucleation in comparison with conventional laparoscopic partial nephrectomy in the treatment of T1a renal cell carcinoma.

DETAILED DESCRIPTION:
Microwave ablation has been widely used in the minimally-invasive treatment of renal tumors. Recently, a technique of laparoscopic microwave ablation-assisted renal tumor enucleation was developed, but the experience was preliminary. This study aims to evaluate the feasibility, safety and efficiency of this technique, particularly its role in the preservation of renal function, in comparison with conventional laparoscopic partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients with sporadic, unilateral, newly diagnosed T1a presumed renal cell carcinoma
* exophytic cancer
* distance from the hilar renal vessels and urinary collecting system >= 1cm
* patients with normal contralateral renal function (differential renal function of >40% as determined by renal scintigraphy)
* patients giving consent to the participation in the current clinical trial

Exclusion Criteria:

* patients with a history of other renal diseases, such as urinary lithiasis
* patients with a history of renal surgery

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
absolute change in glomerular filtration rate (GFR) of the affected kidney | baseline, 3 months and 12 months
  measured by renal scintigraphy

SECONDARY OUTCOMES:
absolute change in eGFR of the affected kidney | baseline, 3 months, 6 months and 12 months
absolute change in total GFR | baseline and 6 months
  measured by renal scintigraphy
blood loss | during surgery
operation time | during surgery
surgical margin | 1 month
  assessed according to the pathology report of the operation specimen
postoperative complications | up to 6 months
  number of participants with postoperative complications graded by Clavien- Dindo system
progression-free survival | 12 months
local recurrence | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ran Huang, M.D., Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China